CLINICAL TRIAL: NCT04362475
Title: Community Health Through Engagement and Environmental Renewal
Acronym: CHEER
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jeffery Walker, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 300004617
Record Dates: First submitted 2020-04-17; First posted 2020-04-27 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Family Relations; Blight

STUDY DESIGN:
Intervention Model Description: Hypotheses will be tested in a 2 X 2 design that includes the independent and combined effects of two interventions targeting the individual, family, and community level. Participating neighborhoods will be assigned into one of four cells: FYI alone, ESPI alone, FYI and ESPI combined, and Wait List Control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Family Youth Intervention (FYI) (Active Comparator): The primary objective of FYI is to evaluate the effectiveness of a theory-based, peer-supported family strengthening intervention on the primary outcomes in a sample of 120 parent-child pairs living in resource-poor urban neighborhoods in Birmingham. For FYI, we will utilize community health advisors (CHAs) to implement the intervention. CHAs will be recruited from each FYI neighborhood and will be trained in research ethics. CHAs will assist and support FYI participants in mastering the sequential skills of the 12 modules designed to improve maternal, youth, and family functioning. Additionally, CHAs will provide emotional social support that is helpful, hopeful, and trustful.
  Interventions: Behavioral: Community Health through Engagement and Environmental Renewal (CHEER)
- ESPI Environment: Social and Physical Intervention (ESPI) (Active Comparator): ESPI will enroll 500 community members to examine the effect of blight elimination through lot recovery on primary outcomes of improved social interaction, social cohesion around common neighborhood norms, and collective efficacy to effect change in the neighborhoods . Neighborhood residents will select a cluster of lots (2-3) for lot recovery that are highly visible in the neighborhood (e.g. on a main thoroughfare). The community residents will lead the neighborhood projects. In some cases, neighborhood residents will personally undertake all or part of the greening projects.
  Interventions: Behavioral: Community Health through Engagement and Environmental Renewal (CHEER)
- Wait-List Control (Other): The two communities will get ESPI, upon completion of the study.
  Interventions: Behavioral: Community Health through Engagement and Environmental Renewal (CHEER)
- FYI and ESPI (Active Comparator): Two of the eight neighborhoods will receive both FYI and ESPI intervention.
  Interventions: Behavioral: Community Health through Engagement and Environmental Renewal (CHEER)

INTERVENTIONS:
Behavioral: Community Health through Engagement and Environmental Renewal (CHEER) — FYI and ESPI intervention activities will be implemented in the overall study, CHEER. It will also allow us to examine possible synergistic effects of both interventions when implemented in the same neighborhoods. Separate sets of participants will be selected for the FYI comparisons and for the ESPI comparisons. Because the FYI intervention focuses on mothers and their children, participants for the FYI comparisons will be selected by Respondent Driven Sampling of eligible families from the neighborhoods in all four cells. The ESPI intervention targets the whole neighborhood, and thus a random sample of neighborhood residents will be enrolled in each of the four cells. Because the primary outcomes for FYI and ESPI are connected but differ from each other, the FYI samples will be assessed for the FYI outcomes in all four cells and the ESPI samples will be assessed for the ESPI outcomes in all four cells.
  Other Names: Family-Youth Intervention (FYI); ESPI Environment: Social and Physical Intervention (ESPI)

SUMMARY:
Community Health from Engagement and Environmental Renewal (CHEER) will leverage previous Centers for Disease Control and Prevention (CDC) community engagement projects to reach and intervene on a high need population. Disadvantage and poverty have long-term and transgenerational adverse impacts on social interaction and cohesion and residents' emotional and physical health. Mothers living and raising children in these conditions face multiple stressors without the community support previous generations relied on. Decades of research on American cities have connected the social, economic, and physical characteristics of neighborhoods with a lack of social cohesion, inability to maintain shared norms of acceptable behavior,and increases in health disparities and risky behaviors. Social cohesion and collective efficacy inversely associate with depression among youth. In a parallel manner, improved parenting practices and youth behavior directly associate with neighborhood social interactions and social cohesion. While these associations are suggestive, CHEER will directly test causal hypotheses at the neighborhood and family levels in a randomized control trial, that can significantly advance the evidence base for public health interventions: Family Youth Intervention (FYI) and an Environment: Social and Physical Intervention (ESPI) to increase social interaction, social cohesion, and collective efficacy and influence wellbeing of mothers and their youth.

DETAILED DESCRIPTION:
Aim 1 Family System: To test the effect of FYI on primary outcomes of youth psychosocial behaviors and sexual risk compared to a Wait List Control.

1a. FYI will significantly improve our primary outcomes of externalizing (e.g. impulsivity, violence, theft) and internalizing (e.g. depression, withdrawal, anxiety, loneliness) behaviors and early and risky sex (i.e. sexual initiation at less than 16 years of age and sexual intercourse without a condom) (Effectiveness).

1. b. FYI will significantly lower parental stress, improve maternal emotional health, enhance parenting skills and improve youth Social and Emotional Competence (SEC) to change primary outcomes (Mediation).

   Aim 2 Community System: To test the effect of ESPI on neighborhood environment compared to Wait List Control.
2. a. ESPI significantly will increase our primary outcomes of social interaction, social cohesion, collective efficacy, and shared norms compared to wait list control (Effectiveness).

2b. Engaging residents in community-designed and -led projects to develop common spaces will significantly improve neighborhood perceptions (e.g. attractiveness, safety) and provide opportunities for residents to interact to change primary outcomes (Mediation).

Aim 3 Community and Family Systems: To test the effects of combining FYI and ESPI on the same youth and neighborhood environmental outcomes as in Aims 1 and 2 compared to FYI alone, ESPI alone, and a Wait List Control.

3a. ESPI and FYI will significantly reduce primary youth and neighborhood environmental outcomes (Effectiveness).

3b. ESPI and FYI will change neighborhood environmental and family processes to change primary outcomes of adolescent SEC, external and internal behaviors, and early and risky sex (Mediation).

ELIGIBILITY:
Inclusion Criteria:

* For FYI, parents who reside in the FYI intervention neighborhood (North Titusville, South Titusville, Rising -West Princeton, and Belview Heights) and have a child age 11-16 years.
* For ESPI, residents who live in the ESPI intervention neighborhoods (North Titusville, South Titusville, Druid Hills, and Fountain Heights).

Exclusion Criteria:

* For FYI, does not met the above requirements and did not consent to participate.
* For ESPI, not residing in one of the above neighborhoods and did not consent to participate.

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 779 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2024-08-10 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
A change in child behavior using the Child Behavior Checklist | Baseline, 6- and 18-month Follow-up
  The child behavior checklist (CBCL) is the most commonly used tool for assessing emotional and behavioral problems in children. Each item ask how the child feels now or within the past 6 months. Participants choose 2 if the item is very true or often true, circle the 1 if the item is somewhat or sometimes true, and if the item is not true, they circle the 0. There are two broadband scales that combine several of the scales. The internalizing problems score assesses the anxious/depressed, withdrawn/depressed, and somatic complaints score. Externalizing problems cover the rule-breaking and aggressive behavior domains.
Age of sexual initiation | Baseline
  Year of age at sex. Two variables were used to measure sexual initiation. First, adolescents were asked, Have you ever engaged in vaginal intercourse? (0 = no, 1 = yes). In order to capture age of sexual initiation, individuals who indicated that they had engaged in vaginal intercourse were then asked, How old were you the first time this happened? Answer choices ranged continuously from 1 (10 years old) to 9 (18 years or older).
Risky sex | Baseline
  Follow-up questions for individuals endorsing sexual initiation to assess risky sex behavior included reporting the number of lifetime sexual partners, With how many girls (for males)/boys (for females) have you ever had vaginal) intercourse? Please enter the number. Contraceptive use in the last 12 months. Frequency of contraceptive use was also assessed with the following question: In the last 12 months, how often did you or your partner use any method to prevent pregnancy or sexually transmitted disease when you had vaginal sex (NOT including withdrawal or the rhythm method)? Answer choices ranged from 0 (never) to 5 (always).
Project on Human Development in Chicago Neighborhoods: Community Survey- Cohesion Index Subscale | Baseline
  Project on Human Development in Chicago Neighborhoods: Community Survey assesses city-level variables relating to neighborhood structure include how residents define their neighborhoods, how long they have lived in a particular neighborhood, characteristics of their neighborhood, including types of social service agencies available, and if they would consider moving to a different neighborhood and why. Other community variables measure the relationships among neighbors, including how many neighbors a respondent would recognize, how often neighbors socialized, and how often neighbors participated in other activities together. Variables that capture neighborhood social order include respondents' perceptions of neighborhood problems such as litter, graffiti, drinking, drugs, and excessive use of force by police. Respondents were also asked about their normative beliefs regarding violence, money, and various children's behaviors.
Project on Human Development in Chicago Neighborhoods: Community Survey -Control Index | Baseline
  Project on Human Development in Chicago Neighborhoods: Community Survey assesses city-level variables relating to neighborhood structure include how residents define their neighborhoods, how long they have lived in a particular neighborhood, characteristics of their neighborhood, including types of social service agencies available, and if they would consider moving to a different neighborhood and why. Other community variables measure the relationships among neighbors, including how many neighbors a respondent would recognize, how often neighbors socialized, and how often neighbors participated in other activities together. Variables that capture neighborhood social order include respondents' perceptions of neighborhood problems such as litter, graffiti, drinking, drugs, and excessive use of force by police. Respondents were also asked about their normative beliefs regarding violence, money, and various children's behaviors.
Project on Human Development in Chicago Neighborhoods: Community Survey- Dev13yr index | Baseline
  Project on Human Development in Chicago Neighborhoods: Community Survey assesses city-level variables relating to neighborhood structure include how residents define their neighborhoods, how long they have lived in a particular neighborhood, characteristics of their neighborhood, including types of social service agencies available, and if they would consider moving to a different neighborhood and why. Other community variables measure the relationships among neighbors, including how many neighbors a respondent would recognize, how often neighbors socialized, and how often neighbors participated in other activities together. Variables that capture neighborhood social order include respondents' perceptions of neighborhood problems such as litter, graffiti, drinking, drugs, and excessive use of force by police. Respondents were also asked about their normative beliefs regarding violence, money, and various children's behaviors.
Social Contacts and Resources Scale | Baseline
  Social Contacts and Resources Scale, a 5-item measure of social activities with their neighbors (e.g., How often do you and other people in your neighborhood visit in each other's homes or on the street?) (Donald and Ware 1982). Responses ranged from 1 (never) to 4 (often). Items were averaged to derive a total score with higher scores indicating greater social resources.

SECONDARY OUTCOMES:
A change in emotional competence using the Social Emotional Competence Questionnaire | Baseline, 6- and 18-month Follow-up
  The Social-Emotional Competence Questionnaire (SECQ) is a survey designed to assess how children and adolescents (grades 3 to 12) are aware of themselves as well as others and how they respond to the contexts of family, school, and community personally, socially and ethically. The 25-item questionnaire is answered on a likert scale.
A change in communication using the Parent-child communication | Baseline, 6- and 18-month Follow-up
  Parent-Adolescent Communication Scale (Barnes & Olson, 1982). The scale is composed of 20 items that measure the degree of openness and lack of problems in family communication. Items in the scale were developed with multiple referents such as "my child,""my parent," making it applicable to both parent and child perspectives. For example, an item on the child version that reads "It is very easy for me to express all of my true feelings to my parent," appears as "It is very easy for me to express all of my true feelings to my child" on the parent version. Response options were on a 5-point Likert scale (1 = strongly disagree, 5 = strongly agree).
A change is parental nurturance using the Parental Nurturance Scale | Baseline, 6- and 18-month Follow-up
  Parental Nurturance Scale, a 24-item Likert-type scale used to measure parental nurturance from the point of view of an individual evaluating the nurturance he or she received from their parents. Examples of items from the Mother's Nurturance Scale are: "My mother seldom says nice things about me," "My mother is often critical of me and nothing I ever do seems to please her," and "My mother enjoys spending time with me."
A change in family functioning using the Family Assessment Device | Baseline, 6- and 18-month Follow-up
  Family Assessment Device (FAD) measures structural, organizational, and transactional characteristics of families. It consists of 6 scales that assess the 6 dimensions- affective involvement, affective responsiveness, behavioral control, communication, problem solving, and roles - as well as a 7th scale measuring general family functioning. The measure is comprised of 60 statements about a family; respondents (typically, all family members ages 12+) are asked to rate how well each statement describes their own family. The FAD is scored by adding the responses (1-4) for each scale and dividing by the number of items in each scale (6-12). Higher scores indicate worse levels of family functioning.
A change in coping with stress using the Cohen Perceived Stress Scale | Baseline, 6- and 18-month Follow-up
  The Perceived Stress Scale (PSS) is the most widely used psychological instrument for measuring the perception of stress. It is a measure of the degree to which situations in one's life are appraised as stressful. Items were designed to tap how unpredictable, uncontrollable, and overloaded respondents find their lives. The questions in the PSS ask about feelings and thoughts during the last month. In each case, respondents are asked how often they felt a certain way. PSS scores are obtained by reversing responses (e.g., 0 = 4, 1 = 3, 2 = 2, 3 = 1 & 4 = 0) to the four positively stated items (items 4, 5, 7, & 8) and then summing across all scale items. A short 4 item scale can be made from questions 2, 4, 5 and 10 of the PSS 10 item scale.
A change in coping using the Coping Self-Efficacy Scale | Baseline, 6- and 18-month Follow-up
  Coping Self-Efficacy (CSE) was assessed with a 26-item measure of perceived self-efficacy for coping with challenges and threats. Participants are asked, 'When things aren't going well for you, or when you're having problems, how confident or certain are you that you can do the following': They were then asked to rate on an 11-point scale the extent to which they believe they could perform behaviors important to adaptive coping, such as 'sort out what can be changed, and what cannot be changed', 'break an upsetting problem down into smaller parts', 'look for something good in a negative situation', and 'get emotional support from friends and family'. Anchor points on the scale were 0 ('cannot do at all'), 5 ('moderately certain can do') and 10 ('certain can do'). An overall CSE score was created by summing the item ratings.
A change in resilience using the Connor-Davidson Resilience Scale | Baseline, 6- and 18-month Follow-up
  The Connor-Davidson Resilience scale (CD-RISC) comprises of 25 items, each rated on a 5-point scale (0-4), with higher scores reflecting greater resilience.
A change in depression using The Center for Epidemiologic Studies Depression Scale | Baseline, 6- and 18-month Follow-up
  The Center for Epidemiologic Studies Depression Scale (CES-D) scale is a short self-report scale designed to measure depressive symptomatology in the general population. CES-D is a 20-item scale with responses on a 4-pt Likert with following responses: Rarely or none of the time (less than 1 day), Some or a little of the time (1-2 days), Occasionally or a moderate amount of time (3-4 days), Most or all of the time (5-7 days). CES-D is scored by assigning zeros for answers in the first column, 1 for answers in the second column, 2 for answers in the third column, 3 for answers in the fourth column. The scoring of positive items is reversed. Possible range of scores is zero to 60, with the higher scores indicating the presence of more symptomatology
A change in social support using the Multidimensional Scale of Perceived Social Support | Baseline, 6- and 18-month Follow-up
  The Multidimensional Scale of Perceived Social Support (Zimet et al., 1988) is a 12-item measure of perceived adequacy of social support from three sources: family, friends, & significant other; using a 5-point Likert scale (0 = strongly disagree, 5 = strongly agree).
A change in quality of life using The World Health Organization Quality of Life Brief Scale | Baseline, 6- and 18-month Follow-up
  The World Health Organization Quality of Life Brief Scale (WHOQOL-BREF) is an abbreviated 26-item version which is scored in four domains: Domain 1: Physical health, Domain 2: Psychological, Domain 3: Social relations and Domain 4: Environment. Items inquire 'how much', 'how completely', how often', 'how good' or 'how satisfied' the respondent felt in the last 2 weeks. The scores are transformed on a scale from 0 to 100 to enable comparisons to be made between domains composed of unequal numbers of items.
A change in how parents discipline using the Punitive Discipline Scale | Baseline, 6- and 18-month Follow-up
  Punitive discipline is assessed using four items developed from the "Welfare, Children and Families: A Three-City Study". Parents indicate the frequency of spanking/hitting, scolding, and threatening to spank/hit or threatening to punish. Response categories included 1 = never in past 12 months; 2 = a few times; 3 = once a month or more; 4 = once a week or more; and, 5 = almost everyday.
A change in the level of parental monitoring using the Parental Monitoring Scale | Baseline, 6- and 18-month Follow-up
  An eight-item parental monitoring scale where adolescents reported how often their parents knew where they were and what they were doing after school, on weeknights, and on weekends; they also report whether their parents knew their friends and how often their parents knew if they had completed their homework. All items used a 4-point scale ranging from 1 (almost never), to 2 (sometimes), to 3 (usually), to 4 (almost always). Individual items were averaged to yield a scale score ranging from 1 (low levels of parental monitoring) to 4 (high levels of parental monitoring).
A change in parenting stress using the Parenting Stress Index | Baseline, 6- and 18-month Follow-up
  The Parenting Stress Index Short Form (PSI-SF) is a self-report screening tool that helps providers and families identify the sources and different types of stress that come with parenting. Parents report their level of agreement with 36 items that fall into three subscales: Parental Distress, Difficult Child Characteristics, and Dysfunctional Parent-Child Interaction. Each item is rated on a 5- point Likert scale format, ranged from strongly agree (5) to strongly disagree (1) . The scores were summarized higher raw scores indicate higher levels of stress.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff T Walker, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Center for the Study of Community Health, Birmingham, Alabama, United States

REFERENCES:
- [Background] Collins WJ, Wanamaker MH. Up from slavery? Black intergenerational economic mobility since 1880.
- [Background] National Bureau of Economic Research Working Paper 23395 http://www.nber.org/papers/w23395 (accessed 2018 Jan 27).
- [Background] Shaw CR, McKay HD. Juvenile delinquency and urban areas. Chicago: University of Chicago Press; 1943.
- [Background] Aneshensel CS, Sucoff CA. The neighborhood context of adolescent mental health. J Health Soc Behav. 1996 Dec;37(4):293-310. PMID 8997886
- [Background] Wilson, WJ. The truly disadvantaged. the inner city underclass and public policy. Chicago: University of Chicago Press; 1987.